CLINICAL TRIAL: NCT06367062
Title: A Study of the Effects of General Anesthesia/Surgical Exposure on Distant Cerebral White Matter Development in Children
Brief Title: General Anesthesia/Surgical Exposure on White Matter Development in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2023-T296
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-12

CONDITIONS: Neurodevelopmental Delay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multiple anesthesia group: Children who underwent more than one general anesthesia procedure between the ages of 0-3 years.
  Interventions: Other: MRI
- Single anesthesia group: Children who underwent only one general anesthesia procedure between the ages of 0-3 years.
  Interventions: Other: MRI
- Control group: Children who underwent no general anesthesia procedure between the ages of 0-3 years.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI is used to assess of brain development.

SUMMARY:
International large-scale clinical studies have found that prolonged or repeated exposure to general anesthesia drugs in infancy and early childhood can lead to an increased risk of long-term neurodevelopmental abnormalities in children. The study of neurodevelopmental toxicity of general anesthesia drugs is of great social significance. We have established a rhesus monkey model to study the neurodevelopmental toxicity of general anesthetic drugs, the first time to make a preliminary exploration of the mechanism of myelin developmental toxicity of general anesthetic drugs. Several studies using magnetic resonance scanning found a positive correlation between the number of anesthesia exposures and the maturity of distant brain white matter development in juvenile non-human primates. Clinical evidence for myelin developmental toxicity induced by general anesthetic drugs needs to be collected by conducting multicenter and large-sample clinical studies. Earlier studies have either had low sample sizes, which do not allow for better control of confounding factors; or the study population has been limited to specific disease populations, and the results cannot be extrapolated to normal children. In view of this, based on the applicant's earlier study, this project proposes to recruit children who underwent general anesthesia surgery between 0-3 years of age and are now 12-15 years old; children who did not experience surgery between 0-3 years of age were matched by age-sex to serve as a control group. MRI will be used to assess their brain white matter development, to explore the correlation between anesthesia and anesthesia-related factors and brain white matter development and related neurobehavioral development, and to clarify the effects of anesthesia and surgery on children's brain white matter and related neuropsychological development.

ELIGIBILITY:
Inclusion Criteria:

* Currently between 12 and 15 years of age

Exclusion Criteria:

* Surgical complications such as acute infectious diseases, systemic diseases
* Abnormal findings on cerebral white matter and/or neurobehavioral assessment
* History of neonatal ischemic-hypoxic encephalopathy, bilirubin encephalopathy
* Genetic or chromosomal disorders, neurological disorders (including epilepsy, congenital disorders), or a history of craniocerebral trauma, infectious diseases of the central nervous system, febrile convulsions, congenital heart disease, oncological diseases, and blood disorders
* Autism, attention deficit hyperactivity disorder, or those who have received behavioral therapy and intervention.
* Children with organic damage to the nervous system
* Cardiovascular surgery, neurosurgery or intraoperative hemodynamic instability.

Ages: 12 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Age between 12-15 years.Past history doesn't lead to abnormal brain development.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI-based assessment of brain development | one time, through study completion, an average of 3 month
  Magnetic resonance scanning of T1-weighted images, T2-weighted images, and diffusion tensor imaging (DTI) of both cerebral hemispheres, looking at whole-brain white matter volume as a percentage of total intracranial volume